CLINICAL TRIAL: NCT03832023
Title: Community Intervention for Tuberculosis Active Contact Tracing and Preventive Therapy - a Cluster Randomized Study (CONTACT)
Brief Title: Community-based Tuberculosis Tracing and Preventive Therapy
Acronym: CONTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Epicentre (Other); University of Sheffield (Other); Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Principal Investigator, Maryline Bonnet, Research Director, MD PhD, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0211
Record Dates: First submitted 2019-01-24; First posted 2019-02-06 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Tuberculosis
Keywords: Children; Contact tracing; Preventive therapy; Prophylaxis; Community health workers; Community-based distribution; Standard of care; Screening; Randomized controlled trial; Cameroon; Uganda; Patient outcome assessment
MeSH Terms: conditions — Tuberculosis | interventions — Mass Screening; Residence Characteristics

STUDY DESIGN:
Intervention Model Description: Clusters were selected among facilities participating in the first phase of the CAP-TB project following an initial facility assessment for participating in the CAP-TB project. Facilities with diagnostic and treatment capacity and detecting and minimum of 50 bacteriologically confirmed pulmonary TB cases per year in a rural/semi-rural or semi-urban setting were selected. The facilities correspond to district hospitals in Cameroon and health center IV or district hospitals in Uganda.
  Twenty clusters will be randomized between the intervention and the facility-based model. The randomization unit (cluster) will be the facility where TB cases (index cases) are diagnosed and its catchment area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facility-based model (No Intervention): Standard of care of each country
- Community-based model (Experimental): Screening and initiating preventive therapy in communities
  Interventions: Other: Screening and initiating preventive therapy in communities

INTERVENTIONS:
Other: Screening and initiating preventive therapy in communities — Symptom-based screening of tuberculosis household child contacts by community health workers; initiation of preventive therapy (3 months of a fixed-dose combination of rifampicin-isoniazid or 6 months isoniazid for HIV+ children on protease inhibitors) in the household by a nurse; follow-up of children under preventive therapy by a community health worker for eligible children at community level, and referral of presumptive tuberculosis cases (children and adults) to the facility.
  Arms: Community-based model

SUMMARY:
The many gaps observed in the cascade of care of tuberculosis (TB) child contacts occur mostly in the screening, preventive therapy (PT) initiation and PT completion steps and the main drivers of these gaps are considered to be the health system infrastructure, limited worker resources and parents' reluctance to bring their children to the facility for screening. There would be great advantages of using a symptom-based screening at community level where only the symptomatic contacts are referred to hospital for further evaluation and asymptomatic contacts are started on PT in the community. Household or community-based screening is likely to improve the uptake and acceptability of child contact screening and management as well as adherence to PT and to reduce cost and workload at facility level.

This study proposes to compare the cascade of care between two models for TB screening and management of household TB child contacts in two high TB burden and limited resource countries, Cameroon and Uganda. In the facility-based model, children will be screened at facility (Cameroon) or household level (Uganda) and preventive therapy initiation, refills of PT therapy and follow-up will be done at facility level. In the intervention group (community-based model), child contacts will be screened in the household by a community health worker (CHW). Those with symptoms suggestive of TB will be referred to the facility for TB investigations. Asymptomatic child contacts from high risk groups (under-5 years or HIV infected 5-14) will be initiated on PT (3 months isoniazid-rifampicin) in the household. Refills of PT therapy will also be done in the communities by the CHW. In both models, symptomatic children requiring further investigations for TB diagnosis will be referred to a health facility.

DETAILED DESCRIPTION:
The primary study objective is to compare the proportion of household child TB contacts eligible for PT (under-5 years and HIV-infected children 5-14 years without active TB) who initiate and complete PT using facility-based and decentralized community-based models of care for contact screening and management.

Secondary objectives are:

1. To compare the facility and community-based models in terms of:

   * The full cascade of care for the initiation and completion of PT in child TB contacts < 5 years or HIV+ children 5-14 years .
   * Cascade of care for the detection and treatment of TB in child contacts (all ages):
   * PT tolerability and adherence among eligible child contacts initiated on PT.
   * Treatment uptake and outcomes for child contacts diagnosed with TB .
   * Child contact outcomes at 6 months after enrollment for all child contacts.
   * Acceptability by the parents/guardians, health personnel and community of the different models of care.
   * Cost and cost-effectiveness of the different models.
   * Fidelity of the implementation of the model activities as compared to the protocol.
2. To assess the number of adult contact cases diagnosed with TB through the community-based screening.
3. To compare between the pre- (baseline assessment) and post-intervention (by model of care) data related to:

   * Children diagnosed with TB and registered at facility level and their treatment outcome.
   * Adults diagnosed with TB and registered at facility level and their treatment outcome.
   * PT initiation and outcomes.

This study will be implemented under the frame of the Catalyzing Pediatric TB Innovation (CaP TB) Project, funded by Unitaid and implemented by the Elizabeth Glaser Pediatric AIDS Foundation (EGPAF). The goal of CaP TB is to improve the pediatric TB morbidity and mortality by catalyzing the wide uptake of the new first-line fixed dose combination drugs for children and optimizing the use of these drugs through improved case detection and innovative models of care. In both models of care, contacts with TB suggestive symptoms will be investigated for TB at the cluster facility that is supported by EGPAF within the CaP TB project. In Cameroon the CaP TB project will be implemented in the Central and Littoral regions and in Uganda in the South-West region.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of the index cases

  * Age > 15 years
  * Newly bacteriologically confirmed TB case (less than a month since diagnosis)
  * Reports child contact(s)
  * Written informed consent signed by the index case and by parents/guardians for minors or incapacitated people
* Inclusion of contacts

  * Household contact
  * Age
  * Facility-based model in Cameroon: < 5 years or HIV infected 5-14 years and all self-referred adults or children*.
  * Facility-based model in Uganda and community-based model on both countries: all ages
  * Written informed consent signed by adult contacts and by parents/guardians for minors or incapacitated people
  * Written assent for children > 7 years in Cameroon and ≥8 years in Uganda

Under the facility-based model in Cameroon, although there is no systematic request to screen adults or HIV-negative child contacts 5-14 years old, first inclusions showed that some of them came by themselves for TB screening. This justifies their inclusion in the study in order to ensure the completeness of data for all contacts screened under the facility-based model.

Exclusion Criteria:

- Exclusion of index cases

* Index cases who do not have child household contacts living in the catchment area of one of the study clusters
* Index cases diagnosed with rifampicin resistance, multidrug-resistant (MDR) or extensively drug-resistant (XDR) TB *Index cases from a household screened within the CONTACT study and that does not declare child contacts from another household.*
* Index cases that are prisoners

TB confirmed adult contacts cases living in the same household as an index case already enrolled in the study will not be included as new index cases unless they declare additional contacts from another household

- Exclusion of the contacts

* If the contact is already on PT or on TB treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Completion of preventive therapy | 6 months
  Proportion of child TB contacts <5 years of age and HIV-infected children of 5-14 years of age who initiate and complete the PT of all child contacts <5 years of age and HIV-infected children of 5-14 years of age declared by the index case

SECONDARY OUTCOMES:
Proportion of children screened | 6 months
  Number of children screened among child contacts <5 years or HIV-infected 5-14 years declared by the index case
Proportion of children eligible for PT | 6 months
  Number of children eligible for PT among screened children
Proportion of children started on PT | 6 months
  Number of children started on PT among those eligible for PT
Proportion of children who did not complete PT | 6 months
  Number of children who did not complete PT among those started on PT
Proportion of children with presumptive TB | 1 month
  Number of children with symptoms suggestive of TB among screened children (< 15 years)
Proportion of children investigated for TB | 1 month
  Number of children with presumptive TB investigated for TB
Proportion of children diagnosed with TB | 1 month
  Number of children diagnosed with TB among those with symptoms suggestive of TB
Proportion of children started on TB treatment | 1 month
  Number of children with TB diagnosis who are started on TB treatment
Proportion of adult contacts screened | 1 month
  Number of adult contacts screened among household identified adult contacts
Proportion of adults presumptive TB cases | 1 month
  Number of adults with symptoms suggestive of TB among those screened for TB
Proportion of adults diagnosed with TB | 1 month
  Number of adults presumptive TB cases diagnosed with TB
Proportion of children with serious adverse events | 6 months
  Number of children with serious adverse events among children started on PT
Proportion of children with adverse event of interest | 6 months
  Number of children with adverse event of interest (peripheral neuropathy, clinical hepatotoxicity) among children on PT
Treatment adherence | 6 months
  Ratio of PT dose taken by the child over the total number of doses prescribed
Treatment outcomes of children started on TB treatment | 6 months
  * Cured
  * Treatment completed
  * Failure
  * Death
  * Lost to follow up
  * Transferred out
Proportion of children diagnosed with TB | 6 months
  Number of children diagnosed with TB after initiation of PT or children not initiated on PT and not diagnosed with TB at baseline
TB case detection during pre-intervention period | 2 years
  Number of patients registered in the facility TB register one year before intervention
Proportion of children among all registered TB cases during pre-intervention period | 2 years
  Number of children among all patients diagnosed with TB and registered in the facility TB register one year before intervention
TB treatment outcome of registered TB patients during pre-intervention period | 2 years
  * Cured
  * Treatment completed
  * Failure
  * Death
  * Lost to follow up
  * Transferred out
Number of children started on PT during pre-intervention period | 2 years
  Number of children started on PT from the facility PT register one year before intervention
Completion rate of children started on PT intervention during pre-intervention period | 2 years
  Number of children who completed PT among those started on PT from the facility PT register one year before
Number of household visits by CHW | 2 years
  Number of visits by the CHW to the household for contact screening per household
Proportion of parents/guardians who accept household visit | 2 years
  Acceptability of household visit for contact screening
Reasons of refusal of household visit | 2 years
  Description of screening failures
Preference for household visit versus facility visit | 2 years
  This outcome measures whether the parent/guardian prefers bringing child to the facility rather than having someone coming to his household
Critical events experienced by CHW during household visit | 2 years
  Description of critical events during house visit and how these where dealt with
Transport cost for household visit by CHW | 2 years
  Cost of transportation for the CHW to go from the health facility to a household
Transport cost for parents/guardian for facility-based screening | 2 years
  Cost supported by families to bring child contact to the facility for screening
Time spent to perform household contact screening visit | 2 years
  It includes the time to reach the household, the time spent in the household and the time to go back to the facility for CHW
Proportion of delivered activities compared to the intended activities of the model | 2 years
  This outcome will assess fidelity to study procedures

CONTACTS AND LOCATIONS:
Overall Officials: Boris Tchounga, MD, PHD, Principal Investigator — Elisabeth Glaser Pediatric AIDS Foundation; Daniel Atwine, MD, PhD, Principal Investigator — Epicentre
Locations (25):
- Cameroon (10):
  - Hôpital de district Bonassama, Bonabéri
  - Hôpital de district Log-Baba, Douala
  - Centre Médical d'arrondissement Delangue, Edéa
  - Hôpital de district Mbalmayo, Mbalmayo
  - Hôpital de district Mfou, Mfou
  - Hôpital régional Nkongsamba, Nkongsamba
  - Hôpital de district Okola, Okola
  - Hôpital de district Olembe, Olembé
  - Hôpital de district St Jean de Malte, Penja
  - Hôpital de district Yoko, Yoko
- Uganda (15):
  - Ishongororo HC IV, Ibanda
  - Ruhoko HC IV, Ibanda
  - Kabwohe Clinical Research Center HC II, Kabwohe
  - Kabwohe HC IV, Kabwohe
  - Kitagata Hospital, Kitagata
  - Bubaare HC III, Mbarara
  - Bwizibwera HC IV, Mbarara
  - Kakoba HC III, Mbarara
  - Mbarara Municipal Council HC IV, Mbarara
  - Bwongyera HC III, Ntungamo
  - Itojo Hospital, Ntungamo
  - Kitwe HC IV, Ntungamo
  - Ntungamo Ngoma HC III, Ntungamo
  - Rubaare HC IV, Ntungamo
  - Rwashamaire HC IV, Ntungamo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandalakas AM, Kirchner HL, Walzl G, Gie RP, Schaaf HS, Cotton MF, Grewal HM, Hesseling AC. Optimizing the detection of recent tuberculosis infection in children in a high tuberculosis-HIV burden setting. Am J Respir Crit Care Med. 2015 Apr 1;191(7):820-30. doi: 10.1164/rccm.201406-1165OC. PMID 25622087
- [Background] Rutherford ME, Hill PC, Triasih R, Sinfield R, van Crevel R, Graham SM. Preventive therapy in children exposed to Mycobacterium tuberculosis: problems and solutions. Trop Med Int Health. 2012 Oct;17(10):1264-73. doi: 10.1111/j.1365-3156.2012.03053.x. Epub 2012 Aug 5. PMID 22862994
- [Background] Triasih R, Robertson CF, Duke T, Graham SM. A prospective evaluation of the symptom-based screening approach to the management of children who are contacts of tuberculosis cases. Clin Infect Dis. 2015 Jan 1;60(1):12-8. doi: 10.1093/cid/ciu748. Epub 2014 Sep 30. PMID 25270649
- [Background] Mandalakas AM, Hesseling AC, Gie RP, Schaaf HS, Marais BJ, Sinanovic E. Modelling the cost-effectiveness of strategies to prevent tuberculosis in child contacts in a high-burden setting. Thorax. 2013 Mar;68(3):247-55. doi: 10.1136/thoraxjnl-2011-200933. Epub 2012 Jun 20. PMID 22717944
- [Background] Szkwarko D, Hirsch-Moverman Y, Du Plessis L, Du Preez K, Carr C, Mandalakas AM. Child contact management in high tuberculosis burden countries: A mixed-methods systematic review. PLoS One. 2017 Aug 1;12(8):e0182185. doi: 10.1371/journal.pone.0182185. eCollection 2017. PMID 28763500
- [Background] Graham SM. The management of infection with Mycobacterium tuberculosis in young children post-2015: an opportunity to close the policy-practice gap. Expert Rev Respir Med. 2017 Jan;11(1):41-49. doi: 10.1080/17476348.2016.1267572. Epub 2016 Dec 10. PMID 27910720
- [Background] Egere U, Sillah A, Togun T, Kandeh S, Cole F, Jallow A, Able-Thomas A, Hoelscher M, Heinrich N, Hill PC, Kampmann B. Isoniazid preventive treatment among child contacts of adults with smear-positive tuberculosis in The Gambia. Public Health Action. 2016 Dec 21;6(4):226-231. doi: 10.5588/pha.16.0073. PMID 28123958
- [Derived] Bonnet M, Vasiliu A, Tchounga BK, Cuer B, Fielding K, Ssekyanzi B, Tchakounte Youngui B, Cohn J, Dodd PJ, Tiendrebeogo G, Tchendjou P, Simo L, Okello RF, Kuate Kuate A, Turyahabwe S, Atwine D, Graham SM, Casenghi M; CONTACT study group. Effectiveness of a community-based approach for the investigation and management of children with household tuberculosis contact in Cameroon and Uganda: a cluster-randomised trial. Lancet Glob Health. 2023 Dec;11(12):e1911-e1921. doi: 10.1016/S2214-109X(23)00430-8. Epub 2023 Oct 30. PMID 37918417
- [Derived] Vasiliu A, Tiendrebeogo G, Awolu MM, Akatukwasa C, Tchakounte BY, Ssekyanzi B, Tchounga BK, Atwine D, Casenghi M, Bonnet M; CONTACT study group. Feasibility of a randomized clinical trial evaluating a community intervention for household tuberculosis child contact management in Cameroon and Uganda. Pilot Feasibility Stud. 2022 Feb 11;8(1):39. doi: 10.1186/s40814-022-00996-3. PMID 35148800
- [Derived] Vasiliu A, Eymard-Duvernay S, Tchounga B, Atwine D, de Carvalho E, Ouedraogo S, Kakinda M, Tchendjou P, Turyahabwe S, Kuate AK, Tiendrebeogo G, Dodd PJ, Graham SM, Cohn J, Casenghi M, Bonnet M. Community intervention for child tuberculosis active contact investigation and management: study protocol for a parallel cluster randomized controlled trial. Trials. 2021 Mar 2;22(1):180. doi: 10.1186/s13063-021-05124-9. PMID 33653385